CLINICAL TRIAL: NCT07121075
Title: The Effects of a Dynamic Arm Support in Daily Life. A Mixed Methods Study Including the Different Components of the ICF
Brief Title: The Effects of a Dynamic Arm Support in Daily Life
Status: Recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Focal Meditech BV (Unknown)
Responsible Party: Principal Investigator, Annemie Spooren, Professor Doctor, Hasselt University
Other Study IDs: B1152024000010
Record Dates: First submitted 2025-02-17; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Neuromuscular Disease; Neuromuscular Disability; Assistive Technology; Activities of Daily Living; Occupational Therapy; Upper Limb
Keywords: dynamic arm support; dynamic arm support device; ICF; daily life; outcome measures
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- People with neurological of (neuro)muscular diseases with a dynamic arm support: The cohort consist of individuals who apply for a dynamic arm support at Focal Meditech.
  Interventions: Device: Dynamic arm support

INTERVENTIONS:
Device: Dynamic arm support — The participant will receive a new dynamic arm support.

SUMMARY:
The goal of this mixed method study is to learn about how a dynamic arm support device (DAS) helps people with everyday activities. The study focuses on people with neuro(-muscular) conditions, age 16 and older. The research questions that are formulated, are:

* How does a person experience their daily activities, with and without a DAS?
* What are the contextual (external and personal) factors that influence the use of a DAS?

Participants will take part in three testing sessions. In each session, they must complete a few questionnaires and participate in an interview. The first time, without DAS. In the second and third session, they will be using their DAS (resp. 3 to 4 weeks and 3 months). The data collection will be executed by phone, digital questionnaires and/or paper.

DETAILED DESCRIPTION:
Methodology:

The target group consist of people:

* with neurological of (neuro)muscular diseases
* at the age of 16 years or older
* who are using a dynamic arm support for at least one activity of daily life. This dynamic arm support is developed by Focal Meditech BV (balancer, Flowing, Dowing, Gowing 2 or Top Help)

Study design:

A convergent parallel mixed method study, consisting of a quantitative and a qualitative component will be executed.

Quantitative data will be collected trough various questionnaires and measurements, during three testing sessions. The goal is to include 50 participants (sample size). To make a comparison between daily life with and without a dynamic arm support, paired t-tests or the Wilcoxon signed-rank test will be performed. All tests are two-tailed, with the significance level set at p < 0.05 and a Bonferonni correction. SPSS, version 27.0, will be used for this data analysis.

Qualitative data will be collected trough in-depth interviews. Participant will be recruited through purposive sampling. The number of included participants will be determined by data saturation. Next, data-analysis will be carried out according to a phenomenological hermeneutical method. Analysis will be conducted in NVivo V.12.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 and oler
* Being able to understand and comprehend test instructions
* Using a DAS from Focal Meditech (Balancer, Flowing, Dowing, Gowing 2 or Top Help)

Exclusion Criteria:

/

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals with a neuro(-muscular) or neurological condition who want to use a DAS, and who, after approval of a healthcare provider, also use a DAS.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Test moment 0: Assessment before delivery of dynamic arm support (DAS), Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  The COPM is a semi-structured interview, where the participants give at least 5 activities of daily life. They give a score of satisfaction and performance (between 1 and 10) on these 5 activities.
Psychosocial impact of assistive devices scale (PIADS) | Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  The psychosocial impact of assistive devices scale is a 26-item, self-report questionnaire designed to assess the effects of an assistive device (the DAS) on functional independence, well-being, and quality of life. Scores on competence (between -3 and +3), adaptability (between -3 and +3) and self-esteem (between -3 and +3).

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) - pain | Test moment 0: Assessment before delivery of dynamic arm support (DAS), Test moment1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  The experienced pain, indicated on a VAS scale, between 0 and 10.
The Flow State Scale for Occupational Tasks (FSSOT) | Test moment 0: Assessment before delivery of dynamic arm support (DAS), Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  The Flow State Scale for Occupational Tasks measures flow experiences during an activity with or without a dynamic arm support (DAS). Scores between 0 and 98.
Diary | Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  During a period of 24 hours, participants fill out a diary in which they indicate how often and for what purposes they use their dynamic arm support (DAS).
Caregiver Assistive Technology Outcome Measure (CATOM) | Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  The caregiver Assistive Technology Outcome Measure measures the caregiver's perception of the impacts of dynamic arm support in his or her life.
  Scores between 18 and 90.
In-depth interview | Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  An in-depth interview about:
  * The personal motivation to use the dynamic arm support
  * The external facilitators and barriers
Visual Analogue Scale (VAS) - fatigue | Test moment 0: Assessment before delivery of dynamic arm support (DAS), Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  The experienced fatigue, indicated on a VAS scale. Scores between 0 and 10.
Positive Health | Test moment 0: Assessment before delivery of dynamic arm support (DAS), Test moment 1: assessment 3 weeks after delivery, Test moment 2: assessment 3 months after delivery
  A questionnaire that assesses 6 dimensions: body functions, mental well-being, sense of meaning, quality of life, participation and daily functioning.
  Scores between 0 and 10, on each dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Joke Raats, Doctor, Principal Investigator — UHasselt
Locations (1):
- Focal Meditech BV (their clients in their home situation), Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data will be shared within the responsible investigators and researcher of UHasselt.

REFERENCES:
- [Background] Shank TM, Wee J, Ty J, Rahman T. Quantitative measures with WREX usage. IEEE Int Conf Rehabil Robot. 2017 Jul;2017:1375-1380. doi: 10.1109/ICORR.2017.8009440. PMID 28814012
- [Background] Cruz A, Callaway L, Randall M, Ryan M. Mobile arm supports in Duchenne muscular dystrophy: a pilot study of user experience and outcomes. Disabil Rehabil Assist Technol. 2021 Nov;16(8):880-889. doi: 10.1080/17483107.2020.1749892. Epub 2020 Apr 15. PMID 32293211
- [Background] Coscia M, Cheung VC, Tropea P, Koenig A, Monaco V, Bennis C, Micera S, Bonato P. The effect of arm weight support on upper limb muscle synergies during reaching movements. J Neuroeng Rehabil. 2014 Mar 4;11:22. doi: 10.1186/1743-0003-11-22. PMID 24594139
- [Background] Prange GB, Jannink MJ, Stienen AH, van der Kooij H, Ijzerman MJ, Hermens HJ. Influence of gravity compensation on muscle activation patterns during different temporal phases of arm movements of stroke patients. Neurorehabil Neural Repair. 2009 Jun;23(5):478-85. doi: 10.1177/1545968308328720. Epub 2009 Feb 3. PMID 19190089
- [Background] van der Heide L, de Witte L. The perceived functional benefit of dynamic arm supports in daily life. J Rehabil Res Dev. 2016;53(6):1139-1150. doi: 10.1682/JRRD.2015.06.0099. PMID 28355038
- [Background] Collins, K. M. (2010). Advanced sampling designs in mixed research. Sage handbook of mixed methods in social and behavioral research, 353-377. SAGE Publications, Inc., https://doi.org/10.4135/9781506335193
- [Background] Essers JMN, Murgia A, Peters AA, Janssen MMHP, Meijer K. Recommendations for studies on dynamic arm support devices in people with neuromuscular disorders: a scoping review with expert-based discussion. Disabil Rehabil Assist Technol. 2022 Jul;17(5):487-500. doi: 10.1080/17483107.2020.1806937. Epub 2020 Sep 26. PMID 32981390
- [Background] Essers J, Murgia A, Peters A, Meijer K. Daily Life Benefits and Usage Characteristics of Dynamic Arm Supports in Subjects with Neuromuscular Disorders. Sensors (Basel). 2020 Aug 28;20(17):4864. doi: 10.3390/s20174864. PMID 32872138
- [Background] Lamers I, Cattaneo D, Chen CC, Bertoni R, Van Wijmeersch B, Feys P. Associations of upper limb disability measures on different levels of the International Classification of Functioning, Disability and Health in people with multiple sclerosis. Phys Ther. 2015 Jan;95(1):65-75. doi: 10.2522/ptj.20130588. Epub 2014 Sep 4. PMID 25190063
- [Background] Michielsen ME, Selles RW, Stam HJ, Ribbers GM, Bussmann JB. Quantifying nonuse in chronic stroke patients: a study into paretic, nonparetic, and bimanual upper-limb use in daily life. Arch Phys Med Rehabil. 2012 Nov;93(11):1975-81. doi: 10.1016/j.apmr.2012.03.016. Epub 2012 Mar 28. PMID 22465403
- See also: website of the different types of dynamic arm supports that are used in this study — https://www.focalmeditech.nl/